CLINICAL TRIAL: NCT00949949
Title: Phase I Trial of Everolimus, Gemcitabine, and Cisplatin for Patients With Solid Tumors Refractory to Standard Therapy
Brief Title: Everolimus, Gemcitabine Hydrochloride, and Cisplatin in Treating Patients With Unresectable Solid Tumors Refractory to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0812; NCI-2009-01151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-000809; MC0812 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Cholangiocarcinoma of the Gallbladder; Localized Gallbladder Cancer; Unresectable Gallbladder Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Everolimus; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort I (everolimus and gemcitabine hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and everolimus PO once daily or 3 times weekly.
  Interventions: Drug: everolimus; Drug: gemcitabine hydrochloride
- Cohort II (everolimus, gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 1 hour on days 1 and 8 and everolimus PO once daily or 3 times weekly.
  Interventions: Drug: everolimus; Drug: gemcitabine hydrochloride; Drug: cisplatin
- Cohort III (MTD) (Experimental): Patients receive treatment as in cohort II.
  Interventions: Drug: everolimus; Drug: gemcitabine hydrochloride; Drug: cisplatin

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
  Arms: Cohort II (everolimus, gemcitabine hydrochloride, cisplatin); Cohort III (MTD)

SUMMARY:
This randomized phase I trial is studying the side effects and best dose of everolimus, gemcitabine hydrochloride, and cisplatin in treating patients with unresectable solid tumors refractory to standard therapy. Drugs used in chemotherapy, such as everolimus, gemcitabine hydrochloride, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of concurrently administered everolimus and gemcitabine (gemcitabine hydrochloride) in patients with advanced, refractory solid tumors (two-agent MTD).

II. To determine the maximally tolerated dose of concurrently administered everolimus, gemcitabine and cisplatin in patients with advanced, refractory solid tumors (three-agent MTD).

III. To describe the toxicity of the two treatment combinations. IV. To describe any evidence of the antitumor activity of the two treatment combinations.

V. To obtain pilot data on toxicity and efficacy outcome of everolimus, gemcitabine and cisplatin in patients with cholangiocarcinoma or gallbladder carcinoma. (Cohort III)

OUTLINE: This is a dose-escalation study of gemcitabine hydrochloride and everolimus.

COHORT I: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8 and everolimus orally (PO) once daily or 3 times weekly.

COHORT II: Patients receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 1 hour on days 1 and 8 and everolimus PO once daily or 3 times weekly.

COHORT III: Patients receive treatment as in cohort II.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now unresectable and refractory to or refused all standard treatment for the disease; exception: cancers in which gemcitabine is considered an appropriate initial treatment option
* Cohort III (MTD) Only: Patients with histologic proof of metastatic cholangiocarcinoma or gallbladder carcinoma who have not had previous treatment for metastatic disease or who received gemcitabine >= 6 months ago as part of adjuvant therapy
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet (PLT) >= 100,000/uL
* Total bilirubin =< 1.5 x Institutional upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5x ULN in patients with liver metastases)
* Creatinine =< 1.5 x Institutional ULN
* Alkaline phosphatase =< 5 x Institutional ULN
* Hemoglobin (Hgb) >= 9.0 g/dL
* International normalized ratio (INR) and Partial thromboplastin time (PTT) =< 3.0 x ULN (anticoagulation is allowed if target INR =< 3.0 x ULN on a stable dose of warfarin or on a stable dose of low-molecular-weight [LMW] heparin for > 2 weeks at time of registration)
* Fasting serum glucose < 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN; NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2
* Ability to provide informed consent
* Willingness to return to Mayo Clinic for follow up
* Life expectancy >= 12 weeks
* Women of childbearing potential only: Negative serum pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Clinically significant cardiac disease, especially history of myocardial infarction =< 6 months, or congestive heart failure (New York Heart Association [NYHA] classification III or IV) requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Patients taking strong inhibitors or inducers of CYP3A4
* Prior therapy with everolimus
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to registration
  * Mitomycin C/nitrosoureas =< 6 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biological therapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
  * Radiation to > 25% of bone marrow prior to registration
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* CNS metastases that are not stable for at least 4 weeks prior to registration based on imaging, clinical assessment, and use of steroids
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Current active other malignancy, except non-melanoma skin cancer or carcinoma-in-situ of the cervix
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Severely impaired lung function (i.e., forced expiratory volume in one second [FEV1] < 1 liter)
* Received immunization with attenuated live vaccines =< 7 days prior to study entry or during study period; NOTE: close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus; examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines
* Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C); Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis B virus (HBV) deoxyribonucleic acid (DNA) and hepatitis C virus (HCV) ribonucleic acid (RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Adverse events profile | Up to 3 months post-treatment
  Tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Toxicity profile per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 | Up to 3 months post-treatment
  Defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal Common Toxicity Criteria (CTC) standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
MTD of the combination of everolimus, gemcitabine hydrochloride, and cisplatin | 3 weeks
  Toxicity assessed by NCI CTCAE v3.0.

SECONDARY OUTCOMES:
Response profile | Up to 5 years
  Best response is defined to be the best objective status recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria will be used for tumor evaluation. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Timed endpoints | Up to 5 years
  The data on time-related variables will be summarized descriptively. These include time until any treatment related toxicity, time until treatment related grade 3+ toxicity, time until hematologic nadirs (white blood cells [WBC], ANC, platelets), time to progression and time to treatment failure, where time to treatment failure is defined as the time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Costello, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota